CLINICAL TRIAL: NCT02180763
Title: A Randomized, Cross-over Study to Compare Quality of Life and Satisfaction in Primary Immunodeficient Patients Treated With Subcutaneous Injections of Gammanorm® 165 mg/mL According to the Delivery Device: Injections Using Pump or Rapid Push.
Brief Title: Gammanorm Quality of Life Study in Immunodeficient Patients Using Rapid Push or Pumps
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAN-03
Record Dates: First submitted 2014-06-23; First posted 2014-07-03 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-08

CONDITIONS: Primary Immunodeficiency (PID)
Keywords: Primary Immunodeficiency, PID
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gammanorm® 165 mg/mL (Experimental)
  Interventions: Biological: Gammanorm

INTERVENTIONS:
Biological: Gammanorm — Sub-Q IgG

SUMMARY:
The purpose of this study is to compare satisfaction (LQI questionnaire, factor I: treatment interference) in PID patients receiving subcutaneous injections of Gammanorm® 165 mg/mL according to the delivery device.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years)
* Presenting with primary immunodeficiency
* Having received subcutaneous injections of immunoglobulin at home using an automatic pump for at least 1 month at the time of inclusion
* For whom the investigator decides to maintain immunoglobulin replacement therapy with subcutaneous injections of Gammanorm® 165 mg/mL at home
* Having signed an informed consent form

Exclusion Criteria:

* Patient currently participating in another interventional study at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-04; Primary Completion 2016-08-28 (Actual); Study Completion 2017-08-26 (Actual)

PRIMARY OUTCOMES:
"Life Quality Index" (LQI) score (factor I: treatment interference) | 6 Months
  Primary endpoint for assessment of patient's satisfaction regarding the treatment delivery device (pump or syringe) will be the "Life Quality Index" (LQI) score (factor I: treatment interference) at the end of each 3-month treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Bienvenu, MD, Principal Investigator — Universtiy Hospital of Caen
Locations (8):
- France (8):
  - Haut-Leveque Hospital, Bordeaux
  - University Hospital of Caen, Caen
  - University Hospital of Lille, Lille
  - Hospital Dupuytren, Limoges
  - Clinique Mutualiste, Lyon
  - University Hospital of Reims, Reims
  - University Hospital of Toulouse, Toulouse
  - University Hospital of Tours, Tours

REFERENCES:
- [Derived] Bienvenu B, Cozon G, Mataix Y, Lachaud D, Alix A, Hoarau C, Antier D, Hachulla E, Brice S, Viallard JF, Tamisier S, Fauchais AL, Renon-Carron F, Clerson P, Fardini Y, Crave JC, Miossec P. Rapid Push vs Pump-Infused Subcutaneous Immunoglobulin Treatment: a Randomized Crossover Study of Quality of Life in Primary Immunodeficiency Patients. J Clin Immunol. 2018 May;38(4):503-512. doi: 10.1007/s10875-018-0507-x. Epub 2018 May 31. PMID 29855752